CLINICAL TRIAL: NCT06371092
Title: A Triple-blind Randomized Clinical Trial Comparing the Efficacy of a Desensitizing Agent Used With an At-home Bleaching Technique
Brief Title: Efficacy of a Desensitizing Agent During At-home Bleaching
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Responsible Party: Principal Investigator, Patricia Pereira-Lores, Principal Investigator, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2023/01
Record Dates: First submitted 2024-04-08; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Sensitivity, Tooth
Keywords: Tooth bleaching; Vital bleaching; Desensitizing agents; Tooth sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — UltraEZ

STUDY DESIGN:
Intervention Model Description: Randomized, triple-blind clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- UltraEZ Group (Experimental): Patients put in their bleaching trays the UltraEZ desensitizing gel for 30 minutes before the bleaching treatment every day during three weeks.
  Interventions: Drug: UltraEZ
- Placebo Group (Placebo Comparator): Patients put in their bleaching trays the UltraEZ placebo gel for 30 minutes before the bleaching treatment every day during three weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: UltraEZ — General examination with bite-wings. Dental prophylaxis (dental scaling and polishing with an abrasive paste). Alginate impressions of both arches. Creation of individualized bleaching trays and a position-finder tray of both arches. Application of the UltraEZ gel in the bleaching trays for 30 minutes. Application of the bleaching gel in the bleaching trays during 6-8 hours
  Arms: UltraEZ Group
Drug: Placebo — General examination with bite-wings. Dental prophylaxis (dental scaling and polishing with an abrasive paste). Alginate impressions of both arches. Creation of individualized bleaching trays and a position-finder tray of both arches. Application of the placebo gel in the bleaching trays for 30 minutes. Application of the bleaching gel in the bleaching trays during 6-8 hours
  Arms: Placebo Group

SUMMARY:
The main objective of this study is to evaluate if the use of UltraEZ during at-home bleaching treatment is effective in reducing tooth sensitivity, as well as doesn't affect the degree of tooth bleaching.

DETAILED DESCRIPTION:
1. Visit 1: Study information and delivery of informed consent. Recording of the patient's medical history, general examination, and prophylaxis. Alginate impressions will be taken of the upper and lower arches for all patients who meet the inclusion criteria. The impressions will be poured into plaster, and individualized bleaching trays will be made for each patient. A positioning guide tray will be fabricated for color measurement.
2. Visit 2: Initial color measurement with a spectrophotometer and the positioning guide. Each patient will receive their individualized trays. Additionally, they will be given 3 syringes of bleaching agent (Opalescence 16%, Ultradent Products) and one syringe of desensitizing agent (UltraEZ, Ultradent Products) or placebo (glycerin), according to their study group. Both the desensitizing agent and placebo will be dispensed in identical syringes, coded as A and B, to ensure the blinding of the study; only the clinician responsible for randomization knows the coding. Each patient will be provided with an instruction sheet and recording sheets to fill out daily during the 3-week study period. They will record the degree of dental sensitivity .
3. Visit 3: First-week bleaching review. Data collection (color + sensitivity).
4. Visit 4: Second-week bleaching review. Data collection (color + sensitivity).
5. Visit 5: Third-week bleaching review and end of the study. Data collection (color + sensitivity).

ELIGIBILITY:
Inclusion Criteria:

* No oral or systemic pathology
* Periodontally healthy
* No cavities
* Tooth shade of the upper and lower canines A2 or darker

Exclusion Criteria:

* Adhesive restorations or prostheses in the anterior region
* Enamel or dentin alterations
* Smoking
* Pregnant women
* Undergone prior bleaching treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Questionnaire of dental sensitivity | Daily, during 3 weeks
  Patients should answer a dental sensitivity questionnaire. A a 5-point subjective numerical classification scale will be used (0=no sensitivity, 1=light, 2=mild, 3=considerable and 4=severe). Patients will a score of 0 during the treatment will be defined as patients with no sensitivity. The individual highest recorded score will be the grade of intensity for each patient.

SECONDARY OUTCOMES:
Shade evaluation with a dental spectrophotometer | Once a week, during 3 weeks
  The color will be measured with a dental spectrophotometer and the parameters L (Lightness), C (Chroma) and H (Hue) will be recorded. To determine the color change between visits the CIEDE2000 formula will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Medicine and Dentistry, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No